CLINICAL TRIAL: NCT06380842
Title: Organ Dysfunction Change in Acute Necrotizing Pancreatitis Patients With Sepsis Undergoing Open Necrosectomy
Brief Title: Organ Dysfunction Change in Acute Necrotizing Pancreatitis Patients With Sepsis After Open Necrosectomy
Status: Recruiting | Type: Observational
Sponsor: Chunling Jiang (Other)
Responsible Party: Sponsor-Investigator, Chunling Jiang, Professor, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: 2023HX1970
Record Dates: First submitted 2024-03-26; First posted 2024-04-24 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Necrotizing Pancreatitis
Keywords: Acute Necrotizing Pancreatitis; sepsis; organ dysfunction
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pancreatitis with sepsis patients' organ dysfunction progression after open necrosectomy: Acute necrotizing pancreatitis patients with sepsis undergoing open necrosectomy will be measured SOFA scores at a special time point to characterize organ dysfunction experience profiles.
  Interventions: Other: Necrotizing Pancreatitis patients' organ dysfunction progression

INTERVENTIONS:
Other: Necrotizing Pancreatitis patients' organ dysfunction progression — Study the dynamic nature of organ dysfunction

SUMMARY:
The purpose of this study is to characterize organ dysfunction change in acute necrotizing pancreatitis patients with sepsis after open necrosectomy.

DETAILED DESCRIPTION:
Before surgery, study participants will be asked questions about age, gender, education level, etc. Study participants will also be questioned regarding pancreatic symptoms, as measured on the patient-Reported Outcome Scale in Acute Pancreatitis (including, pain, abdominal distention, eating, bowel movements, nausea and vomiting, thirst, and weakness). Organ dysfunction was defined according to the sequential organ failure assessment (SOFA) score. The SOFA score will be measured at preoperative (T1), postoperative day 1 (T2), postoperative day 3 (T3), postoperative day 7, or at hospital discharge, whichever comes first (T4). Following discharge from the hospital, study participants will be contacted at 1 month, 3 months, 6 months, and 1 year after surgery, and asked to complete a survey about their pancreatic symptoms and survival status after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older
2. Diagnosis of Acute pancreatitis according to the revised Atlanta classification, requires two of the following three criteria: (A) typical abdominal pain, (B) an increase in serum amylase or lipase levels higher than three times the upper limit of normality, and (C) signs of AP in imaging
3. Patients with confirmed or suspected infected pancreatic or peripancreatic necrosis were scheduled for open necrosectomy
4. Meet Sepsis-3 criteria

Exclusion Criteria:

1. Patients refuse to participate
2. Patients undergo repeat surgery on the same site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute necrotizing pancreatitis Patients with sepsis scheduled for open necrosectomy will be invited to participate in this study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Measure organ dysfunction change after open necrosectomy with respect to time | up to postoperative day 7, or at hospital discharge, whichever comes first
  Organ dysfunction will be measured using sequential organ failure assessment score scale. The scores range from 0 (normal) to 4(most abnormal) for each organ, with higher scores indicating worse health status

SECONDARY OUTCOMES:
incidence of a composite of major complications | up to postoperative day 28
  Major complications were defined as new-onset organ failure (ie, cardiovascular, pulmonary, or renal)
Incidence of ICU mortality | through study completion, an average of 1year
  Death occurred in ICU
Incidence of hospital mortality | through study completion, an average of 1 year
  Death occurred in hospital
Incidence of 28-day mortality | through study completion, an average of 1 year
  Death occurred within 28-day after surgery
Incidence of one year mortality | through study completion, an average of 1 year
  Death occurred within one year after surgery
ICU length of hospital stay | through study completion, an average of 1 year
  Determined by the number of days from ICU admittance to discharge from ICU
Length of hospital stay | through study completion，an average of 1 year
  Determined by the number of days from admittance to discharge
The pancreatic symptoms score | up to 1 year
  Pancreatic symptom scores will be measured at preoperative, postoperative day 1, day 2, day 3, day 7, or at hospital discharge, whichever comes first, at 1 month, 3 months, 6 months, and 1 year postoperatively. Both were measured using the Patient-Reported Outcome Scale, which ranges from 0 to 10 for each symptom; The overall range is from 0 to 70, with higher scores indicating higher symptom intensity.
The levels of inflammatory factor CRP | preoperative, postoperative day 1, day 3 and day 7 or at hospital discharge, whichever came first.
  Peripheral blood CRP
The levels of inflammatory cytokines IL-6 | preoperative, postoperative day 1, day 3 and day 7 or at hospital discharge, whichever came first.
  cytokines IL-6
The levels of inflammatory procalcitonin | preoperative, postoperative day 1, day 3 and day 7 or at hospital discharge, whichever came first.
  procalcitonin was measured at preoperative, postoperative day 1, day 3 and day 7 or at hospital discharge, whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Fengming Luo, PhD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, China, China

IPD SHARING:
Plan to Share IPD: No